CLINICAL TRIAL: NCT01015495
Title: Ranibizumab Therapy for Choroidal Neovascularization Associated With Angioid Streaks
Brief Title: Ranibizumab Therapy for Choroidal Neovascularization (CNV) Asociated With Angioid Streaks
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Not enough patients within the time frame to allow for a meaningful study.
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Jennifer I. Lim, Professor of Ophthalmology, Director of Retina Services, Department of Ophthalmology and Visual Sciences, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fvf 3763s
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Angioid Streaks
Keywords: angioid streaks; CNV; intra vitreal ranibizumab
MeSH Terms: conditions — Angioid Streaks | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ranibizumab (Experimental)
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — 0.5 mg dose of ranibizumab. Treatment will be given at baseline, month 1, and month 2, and then monthly until OCT shows absence of subretinal fluid and FA shows absence of leakage
  Other Names: Lucentis

SUMMARY:
The purpose of this study is to determine whether injections of ranibizumab into the eye are safe and well tolerated when given to subjects in multiple doses.

DETAILED DESCRIPTION:
Choroidal neovascularization is a hallmark of angioid streaks, and presumably VEGF-driven. Ranibizumab has been shown to be effective in CNV secondary to age-related macular degeneration. Therefore, we hypothesize that ranibizumab may be efficacious in the treatment of CNV secondary to angioid streaks

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Angioid streaks
* Subfoveal CNV of recent onset with the following characteristics
* Absence of subfoveal fibrosis
* Fibrosis less than 25% of the lesion
* Presence of blood, subretinal fluid, and/or lipid
* New onset symptoms within 12 weeks
* Visual acuity 20/40 to 20/800 on an ETDRS chart

Exclusion Criteria:

* Prior treatment of subfoveal CNV in the study eye
* Age-related macular degeneration
* Uncontrolled glaucoma
* High myopia (> -10.00 D spherical equivalent)
* Prior retinal detachment
* Media opacity preventing adequate view of the retina
* Planned cataract surgery in the next 3 months
* Current chemotherapy for cancer
* Immunocompromised state
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* History of any previous treatment for angioid streaks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures for safety and tolerability are the following: • Incidence and severity of ocular adverse events, as identified by eye examination (including visual acuity testing) | Month 12

SECONDARY OUTCOMES:
Proportion of patients that lose fewer than 15 letters from baseline at months 6 and 12 as assessed by the number of letters read correctly on the ETDRS eye chart at a starting test distance of 4 meters at months 6 and 12 | Month 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer I Lim, MD, Principal Investigator — UIC Eye and Ear Infirmary

REFERENCES:
- See also: UIC-Ophthalmology home page — http://www.uic.edu/com/eye/